CLINICAL TRIAL: NCT01031134
Title: Shared Decision-Making for Elderly Depressed Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH084872-01A1 (NIH); 1R01MH084872-01A1 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shared Decision Making (Experimental): 1 in person session followed by 2 telephone calls 1 and 2 weeks later.
  Interventions: Behavioral: Shared Decision Making
- Usual Care (Active Comparator): Physician Usual Care of depressed patients.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Shared Decision Making — Shared decision-making, in contrast to traditional medical decision-making, involves a collaborative process where patients discuss personal values and preferences and clinicians provide information to arrive at an agreed upon treatment decision. The focus of the intervention is to empower elderly depressed primary care patients and help them efficiently arrive at a treatment decision that can be successfully implemented.
  Arms: Shared Decision Making
Other: Usual Care — Usual Care reflects the standard of care in primary care practice: following physician recommendation for treatment. Physicians will recommend some form of depression treatment. This may take the form of an antidepressant prescription or psychotherapy referral. The physician will encourage patients to telephone with any questions. Following the treatment recommendation provided to the patient, the physician will provide care as usual.
  Arms: Usual Care

SUMMARY:
Shared decision-making (SDM), in contrast to traditional medical decision-making, involves a collaborative process where patients discuss personal values and preferences and clinicians provide information to arrive at an agreed upon treatment decision. The proposed study will evaluate the impact of a brief SDM nursing intervention among elderly, depressed primary care patient subjects in comparison to physician recommended Usual Care. The focus of the SDM intervention is to empower depressed patients and help them arrive at a treatment decision that can be successfully carried out.

DETAILED DESCRIPTION:
Shared Decision Making (SDM) may be particularly relevant for depressed individuals, as it seeks to enhance their autonomy and empowerment in a manner that directly addresses the helplessness and hopelessness associated with depression. Shared decision-making interventions are being developed for depression in primary care, but have yet to be adequately tested. It is also unknown whether the same premises regarding shared decision-making's ability to enhance autonomy and empowerment pertain to elderly populations.

This randomized study will recruit elderly depressed primary care patient subjects and evaluate the impact of a three-session SDM nursing intervention on their (1) adherence to antidepressant medication or psychotherapy and on (2) their reduction in depressive symptoms. The comparison group will be physician-recommended Usual Care (UC). The focus of the SDM intervention is to empower elderly depressed primary care patients and help them efficiently arrive at a treatment decision that can be successfully implemented.

The study randomizes physicians to provide their depressed patients with SDM or UC. A total of 210 elderly depressed patient subjects whose physicians recommend starting depression treatment, will receive either Shared Decision-Making (SDM) or the physician recommended Usual Care (UC) comparison condition. Participants will be assessed at baseline and at weeks 4, 8, 12, and 24 to determine treatment adherence and depressive status. Nurses currently employed by the participating physicians will administer the SDM intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years and older;
* Medical outpatient presenting to Lincoln Hospital, Bronx NY, the New York City Health and Hospitals Corporation (HHC);
* Screen positive (PHQ-9 score>9 for depression, in addition to primary care physician recommendation for depression treatment.

Exclusion Criteria:

* Presence of significant alcohol or substance abuse, psychotic disorder, or bipolar disorder;
* High suicide risk, i.e. intent or plan to attempt suicide in near future;
* Current treatment with antidepressant medication or psychotherapy prior to index physician visit (with the exception of low doses of antidepressant medication for pain disorders);
* Cognitive impairment: MMSE score <20 or clinical diagnosis of dementia;
* Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver, or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs often causing depression, e.g., steroids, reserpine, alpha-methyl-dopa, tamoxifen, vincristine;
* Aphasia interfering with communication.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Raue, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Lincoln Hospital - the New York City Health and Hospitals Corporation (HHC), The Bronx, New York
  - Cornell Institute of Geriatric Psychiatry, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raue PJ, Schulberg HC, Bruce ML, Banerjee S, Artis A, Espejo M, Catalan I, Romero S. Effectiveness of Shared Decision-Making for Elderly Depressed Minority Primary Care Patients. Am J Geriatr Psychiatry. 2019 Aug;27(8):883-893. doi: 10.1016/j.jagp.2019.02.016. Epub 2019 Mar 1. PMID 30967321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shared Decision Making | Usual Care
Started | 114 | 88
Completed | 103 | 78
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shared Decision Making | Usual Care | Total
Number analyzed (Participants) | 114 | 88 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 114 | 88 | 202
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 72 | 164
  Male | 22 | 16 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 83 | 184
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 25 | 59
  White | 58 | 53 | 111
  More than one race | 22 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 88 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Adhered to Physician Recommended Treatment
Description: Any mental health service use over 12 weeks.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Shared Decision Making | Usual Care
Number analyzed (Participants) | 103 | 78
Participants | 40 | 16

2. Secondary Outcome: Change in Hamilton Depression Rating Scale Scores
Description: Hamilton Depression Rating Scale change score from baseline to 12 weeks. This scale measures severity of depressive symptoms (range 0-76), with higher scores indicating more severe symptomatology.
Time Frame: Baseline and 12 week
Population: fewer number of participants in comparison to primary outcome measure reflect greater numbers of missing observations for the Hamilton outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shared Decision Making | Usual Care
Number analyzed (Participants) | 84 | 66
units on a scale | -6.05 (7.03) | -7.35 (6.97)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Shared Decision Making | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/114 | 0/88
Serious Adverse Events (participants affected / at risk) | 49/114 | 47/88
Other Adverse Events (participants affected / at risk) | 0/114 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Shared Decision Making (N=114) | Usual Care (N=88)
ER visit (General disorders) | 21 | 21
hospitalization (Surgical and medical procedures) | 1 | 1
hospitalization (Gastrointestinal disorders) | 0 | 1
hospitalization (General disorders) | 0 | 2
ambulatory surgery (Surgical and medical procedures) | 2 | 0
ER visit (Cardiac disorders) | 4 | 9
ER visit (Gastrointestinal disorders) | 1 | 0
ER visit (Infections and infestations) | 2 | 2
ER visit (Injury, poisoning and procedural complications) | 2 | 3
ER visit (Psychiatric disorders) | 1 | 3
ER visit (Renal and urinary disorders) | 1 | 0
ER visit (Respiratory, thoracic and mediastinal disorders) | 6 | 3
ER visit (Surgical and medical procedures) | 1 | 0
ER visit (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No